CLINICAL TRIAL: NCT06431997
Title: Effects of Time-restricted Eating on the Incidence of Gestational Diabetes Mellitus in High-risk Populations: a Randomized Controlled Study
Brief Title: A Study of the Intervention of Time-restricted Eating in High-risk Populations of GDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shenzhen Maternity & Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Yu Xiong, Clinical Professor, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FD153502
Record Dates: First submitted 2024-04-23; First posted 2024-05-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-04

CONDITIONS: Gestational Diabetes Mellitus; Dietary Habits; Lifestyle Intervention; Randomized Controlled Study
Keywords: Gestational Diabetes Mellitus; Metabolic Diseases
MeSH Terms: conditions — Diabetes, Gestational; Feeding Behavior; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRE(Time-restricted eating group) (Experimental): Participants assigned to the TRE group will be instructed to consume prescribed calories in a 10-hour eating window (from 8:30 am to 18:30 pm) each day and only noncaloric beverages were permitted outside of the eating window over 3 months (from 14-26 gestational weeks).
  Interventions: Behavioral: Time-limited eating
- SOC (standard of care group) (No Intervention): Participants in the SOC group will be instructed to consume prescribed calories following habitual daily eating schedule over 3 months.

INTERVENTIONS:
Behavioral: Time-limited eating — All participants will be instructed to follow a diet of 1800-2200 kcal/d (45-50% of energy from carbohydrate, 15-20% from protein, 25-30% from fat) based primarily on Dietary Guidelines for Chinese Residents (2022), Dietary guidelines for pregnant women and Guideline of Diagnosis and Treatment of Hyperglycemia in Pregnancy (2022). Participants assigned to the TRE group will be instructed to consume prescribed calories in a 10-hour eating window (from 8:30 am to 18:30 pm) each day and only noncaloric beverages were permitted outside of the eating window over 3 months (from 14-26 gestational weeks). Participants in the SOC group will be instructed to consume prescribed calories following habitual daily eating schedule over 3 months.
  Arms: TRE(Time-restricted eating group)

SUMMARY:
This is a randomized controlled trial, aiming to investigate whether a time-restricted eating (TRE) can reduce the incidence of gestational diabetes mellitus (GDM) in high-risk pregnant women. Investigators intend to conduct a 3-month randomized controlled study to compare the effects of 10-hour TRE and habitual eating time on GDM .

DETAILED DESCRIPTION:
Investigators present a multicenter, open-label and parallel-group randomized study. Total 240 women in early pregnancy were randomly assigned to TRE group and SOC (standard of care) group according to the ratio of 1: 1. Participants assigned to the TRE group will be instructed to consume prescribed calories in a 10-hour eating window (from 8:30 am to 18:30 pm) each day and only noncaloric beverages were permitted outside of the eating window over 3 months (from 14-26 gestational weeks). Participants in the SOC group will be instructed to consume prescribed calories following habitual daily eating schedule over 3 months. All participants should follow moderate-intensity physical activity for about 30 minutes every day, and receive diet and exercise counseling during the study period. GDM was diagnosed by 75g oral glucose tolerance test (OGTT) test at about 26 gestational weeks.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-50 years;
2. The risk for GDM includes overweight or obesity (BMI ≥ 24 kg/m2 before pregnancy), first-degree relative with diabetes, history of cardiovascular disease, hypertension (≥130/80 mmHg or on therapy for hypertension), HDL cholesterol level < 1 mmol/L and/or a triglyceride level > 2.8 mmol/L, history of GDM, history of macrosomia delivery, individuals with polycystic ovary syndrome, repeated positive fasting urine glucose in the first trimester, or age>45 years according to Guideline of Diagnosis and Treatment of Hyperglycemia in Pregnancy (2022);
3. Less than 14 weeks of gestation;
4. Able to read and complete questionnaires in Chinese;
5. singleton pregnancy.

Exclusion criteria:

1. Pregestational diabetes (including diabetes diagnosed before conception; fasting blood glucose ≥ 7.0 mmol/L or HbA1c ≥ 6.5% in the first trimester; typical symptoms of hyperglycemia or hyperglycemic crisis with optional blood glucose ≥ 11.1 mmol/L);
2. Impaired glucose tolerance (including fasting blood glucose ≥ 5.6 mmol/L or two fasting blood glucose ≥ 5.1 mmol/L in the first trimester);
3. Current or recent use of drugs that affect glucose metabolism such as metformin, glucocorticoids and Orlistat;
4. Severe comorbidities (including cardiac diseases, kidney diseases, hepatopathy, autoimmune diseases, uncontrolled thyroid disease, previous or current malignant tumors, etc.);
5. Fetal malformations or chromosomal abnormalities;
6. Cervical insufficiency (including ultrasonic cervical length < 25 mm before 24 weeks of gestation, history of spontaneous preterm birth at 14-36 weeks of previous pregnancy, or cervical dilation in the past or current pregnancy);
7. Exercise contraindications (including continuous vaginal bleeding, threatened premature labor, placenta previa, premature rupture of membranes, severe anemia, etc.);
8. Drug abuse, which refers to the repetitive, heavy use of drugs with dependent characteristics such as narcotic, psychotropic substances, tobacco and alcohol;
9. Hyperemesis gravidarum, which refers to the severe and persistent nausea and vomiting, unable to eat or eat little that leads to dehydration, ketosis and even acidosis;
10. On a special or prescribed diet for other reasons;
11. Eating window<10 h.

Exit criteria：

1. Failure to comply with or assume the corresponding responsibilities and obligations of the informed agreement;
2. Pregnant women who terminate their pregnancy before completing GDM diagnosis and screening at 24-28 weeks of pregnancy will automatically withdraw from the group, such as severe fetal malformation, eclampsia, abortion, etc.
3. Major diseases, such as particularly serious obstetric medical events, malignant tumors, serious cardiovascular and cerebrovascular diseases, brain injuries, paralysis and other major diseases, can not continue to accept this intervention plan and follow-up, and withdraw from the study;
4. Accidental disability or death caused by non-intervention factors occurred during the study period, and he withdrew from the study;
5. Subjects are subjectively unwilling to continue to accept the intervention program, and sign the withdrawal agreement to withdraw from the group on a voluntary basis, and decide whether to continue to follow up the pregnancy process and outcome according to the specific contents of the withdrawal statement.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of GDM | 26 gestational weeks
  Diagnosed by the 75g oral glucose tolerance test (OGTT).

SECONDARY OUTCOMES:
Number of newborns with macrosomia | At delivery
  Number of newborns with birth weight ≥4000g.
Number of newborns with low birth weight | At delivery
  Number of newborns with birth weight <2500g.
Number of newborns large for gestational age (LGA) | At delivery
  Number of newborns with weight lies above the 90th percentile for the gestational age.
Number of newborns small for gestational age (SGA) | At delivery
  Number of newborns with weight lies below the 10th percentile for the gestational age.
Incidence of shoulder dystocia | At delivery
  The incidence of the condition in which normal traction on the fetal head does not lead to the delivery of the shoulders.
Number of newborns with birth injury | At delivery
  Number of newborns with an impairment of the neonate's body function or structure due to an adverse event that occurred at birth.
Number of neonatus with neonatal intensive care unit (NICU) admission | Within the first 28 days after delivery
  Number of neonatus with neonatal intensive care unit (NICU) admission.
Number of neonatus with neonatal respiratory distress | Within the first 28 days after delivery
  Number of neonatus with clinical symptoms including tachypnea, nasal flaring, grunting, retractions (subcostal, intercostal, supracostal, jugular), cyanosis, apnea, bradypnea, irregular breathing, inspiratory stridor, wheeze and hypoxia, etc.
Number of neonatus with hypoglycemia | Within the first 48 hours after delivery
  Number of neonatus with venous glucose levels <2.6mmol/L.
Number of neonatus with pathologic jaundice | Within the first 28 days after delivery
  Jaundice that arises from factors that alter the usual process involved in bilirubin metabolism in the liver that requires treatment.
Number of neonatus with intraventricular hemorrhage (IVH) of II grade or above | Within the first 28 days after delivery
  Intraventricular hemorrhage (IVH) of II grade or above diagnosed by ultrasound.
Number of neonatus with necrotizing enterocolitis (NEC) | Within the first 28 days after delivery
  Necrotizing enterocolitis (NEC) diagnosed by radiography or surgery.
Number of neonatus managed with assisted ventilation >24 hours via endotracheal tube. | Within 72 hours of birth
  Number of neonatus managed with assisted ventilation >24 hours via endotracheal tube.
Number of neonatus with sepsis. | Within the first 28 days after delivery
  Number of neonatus with septicemia ascertained by blood culture.
The incidence of neonatal death. | Within the first 28 days after delivery
  The incidence of deaths among live births during the first 28 completed days of life.
The level of maternal fasting plasma insulin | at 24-28 gestational weeks
  Maternal fasting plasma insulin level.
The level of maternal HbA1c | at 24-28 gestational weeks
  Maternal venous glycosylated hemoglobin A1c (HbA1c) level.
Insulin resistance calculated by homeostatic model assessment (HOMA-IR) | at 24-28 gestational weeks
  Insulin resistance calculated by homeostatic model assessment (HOMA-IR). HOMA-IR=fasting plasma glucose (FPG)× fasting plasma insulin (FINS)/22.5. The higher HOMA-IR value indicates higher severity of insulin resistance.
Maternal lipid profile | at 24-28 gestational weeks
  Level of maternal venous low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides and total cholesterol.
Maternal change in depression, quality of sleep and quality of life | From pre-pregnancy to 24-28 gestational weeks
  Maternal change in depression, quality of sleep and quality of life measured by the Patient Health Questionnaire-9 (PHQ-9), Pittsburgh sleep quality index (PSQI) and 12-item Short-Form Health Survey Questionnaire (SF-12) according to pre-pregnancy status and 24-28 gestational weeks.
  The Patient Health Questionnaire-9 (PHQ-9): Scores range from 0 to 27, with higher scores indicating severer depression. The standard cut-off score for screening to identify possible major depression is 10 or above.
  Pittsburgh sleep quality index (PSQI): Scores range from 0 to 21, with higher scores indicating worse sleep quality.
  12-item Short-Form Health Survey Questionnaire (SF-12): physical component score (PCS) range from 0 to 100, higher scores are better.
Gestational weight gain | From pre-pregnancy to 24-28 gestational weeks
  Measured according to pre-pregnancy weight and weight at 24-28 gestational weeks.
Change in waist circumference | From pre-pregnancy to 24-28 gestational weeks
  Measured according to pre-pregnancy waist circumference and waist circumference at 24-28 gestational weeks.
Incidence of maternal morbidities | From 24-28 gestational weeks to delivery
  Incidence of hypertensive disorders of pregnancy, hydramnios, placental abruption, preterm/prelabor rupture of membranes (P/PROM), preterm birth, chorioamnionitis, postpartum hemorrhage and still birth.

OTHER OUTCOMES:
Adherence to the intervention | From 14-26 gestational weeks
  Adherence to the intervention measure by Chinese Dietary Guidelines Compliance Index for Pregnant Women (CDGCI-PW) and by counting the number of days in which participants consumed calories outside the time-window or exceeding the upper limit of the required energy intake.
  Chinese Dietary Guidelines Compliance Index for Pregnant Women (CDGCI-PW): Scores range from 0-100, with higher score indicating better adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China